CLINICAL TRIAL: NCT04654507
Title: Efficacy of Corticosteroids in Reducing Renal Scarring in Acute Pyelonephritis in Children:A Multi-centre, Double-blind, Randomized, Placebo-controlled, Clinical Trial
Brief Title: Efficacy of Corticosteroids in Reducing Renal Scarring in Acute Pyelonephritis in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MRC-01-20-085
Record Dates: First submitted 2020-11-30; First posted 2020-12-04 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Urinary Tract Infections in Children; Dexamethasone; Kidney Scarring; Acute Pyelonephritis; Hypertension in Children; Chronic Renal Failure; UTI
MeSH Terms: conditions — Glomerulonephritis; Kidney Failure, Chronic | interventions — Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant dexamethasone (Active Comparator): Drug: Dexamethasone
  Interventions: Drug: Dexamethasone Oral
- Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone Oral — Drug: Dexamethasone 0.3mg/kg/dose twice daily for 3 days
  Other Names: corticosteroids
  Arms: Adjuvant dexamethasone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Urinary tract infection (UTI) is the most frequently occurring serious bacterial infection in young children and accounts 5 to 14% of emergency department visits Formation of renal scarring in children has been associated with serious complications as hypertension, preeclampsia, and end stage renal failure in young age . So, this study aims to determine whether dexamethasone reduces the renal scarring in children will be treated with antibiotics for acute pyelonephritis.

investigators propose to conduct a multi center, randomized, placebo-controlled, double-blind clinical trial, that will evaluate the efficacy of dexamethasone (0.3 mg/kg every 12 hours per day orally for 3 days) in preventing renal scarring in young febrile children (2 months to 14 years) with a first-diagnosed UTI. 120 Participants will be enrolled over a 3-year period from 6 sites.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is the most frequently occurring serious bacterial infection in young children and accounts for 5 to 14% of emergency department visits. UTIs can be divided into asymptomatic bacteriuria, cystitis, and acute pyelonephritis (APN ). The APN is associated with an increased risk of renal damage, acquired through renal scarring. Which is a consequence of the inflammatory and immune response that aim to eradicate the bacteria involved in the UTI.

Parenchymal infection can be solved, but there are a number of poorly understood factors that may perpetuate inflammation, and this would promote the formation of scarring. One of the most relevant factors involved in formation of renal scarring is the production of inflammatory mediators (complement proteins, bactericidal peptides, cytokines , chemokines, ). hence, the use of anti-inflammatory drugs may prevent the release of these mediators and the formation of permanent renal scarring. Renal scarring in childhood has been associated with serious complications as hypertension, preeclampsia, and ESRD in young age.

Current treatment of children with UTI has focused on the treatment of vesicoureteral reflux (VUR) and on the early treatment of UTI with antibiotics. Although the presence of VUR increases the likelihood of bacteria gaining access to the kidney, correction of VUR is not sufficient to prevent scarring. Renal scarring frequently occurs in children who do not have VUR, and early diagnosis and treatment of children with VUR is not associated with a reduction in the incidence of end-stage renal disease. Similarly, early antibiotic therapy is necessary, but it is not sufficient to prevent renal scarring in most children with UTI. Because signs of UTI in children are relatively non-specific, the diagnosis is often delayed. data from many studies have shown that once the infection has localized to the renal parenchyma, treatment with antibiotics alone does not prevent scarring. hence ,It is clear that the current management is not always effective in preventing renal scarring. The proposed study aims to determine whether dexamethasone therapy - which focuses on modulation of the host inflammatory response - is effective in reducing renal scarring.

ELIGIBILITY:
Inclusion Criteria:

* First episode of acute febrile UTI.
* From 2 months to 14 years of age.
* Fever: ≥ 38.3°C, measured at home or at Pediatric Emergency centers.,

Exclusion Criteria:

* Previous history of UTI.
* Urinary tract abnormalities except VUR.
* Antibiotic use within 7 days of enrollment (except last 48 hours)
* previous renal scarring
* patients included in the study and suffered second pyelonephritis during the first 6 months
* Patients allergic to dexamethasone.
* Endocrinology diseases.
* cancer.
* Planned admission to ICU
* Other bacterial infection as meningitis or pneumonia
* Congenital/acquired immunodeficiency
* Systemic use of corticosteroids or other immunomodulation agents within 14 days of enrollment.

Ages: 2 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Renal scarring comparatively with patients those don't take the medicine | 6 months
  Division of Children With Renal Scarring at the Outcome of (DMSA) Renal Scan [ Time Frame: The outcome DMSA scan will be 6 months from enrollment.] Renal scarring is defined as decreased uptake of tracer with or without loss of contours.
  Three radiologists independently will review all renal DMSA scans for scarring .
  Diagnosis of presence or absence of renal scarring for a kidney , should be endorsed by the majority of readers (2/3).
  The child will be determined to have renal scarring if either kidney or both kidneys have scarring by the majority of readers.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alhandi Omar Helal, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No